CLINICAL TRIAL: NCT02442986
Title: Prospective Observational Study: Comparison of Neurological Outcome in Septic Surgical, Septic Non-surgical and Non-septic Patients on ICU
Brief Title: Neurological Outcome in Surgical and Non-surgical Septic Patients
Acronym: NOSEPP
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, MD, University of Rostock
Other Study IDs: URostock
Record Dates: First submitted 2015-04-29; First posted 2015-05-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Critical-Illness; Polyneuropathy; Myopathy; Septic Encephalopathy
Keywords: weaning failure; polyneuropathy; encephalopathy; sepsis
MeSH Terms: conditions — Critical Illness; Polyneuropathies; Muscular Diseases; Sepsis-Associated Encephalopathy; Brain Diseases; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Septic Shock or severe sepsis: Septic patients on ICU with severe sepsis or septic shock.
- Non-Septic, Surgical Patients: Non-septic patients after surgical treatment and anesthesia on ICU.
- Non-Septic, Non-Surgical Patients: Patients without sepsis criteria treated on ICU, non-surgical patients.

SUMMARY:
Systemic inflammation and sepsis cause multi organ failure including severe neurologic impairment in the course of disease. Neurologic failure typically presents as critical-illness-polyneuropathy/-myopathy and septic encephalopathy during sepsis and is associated with an increased mortality rate.

Clinical parameters to determine the neurologic entities during the course of sepsis are heterogeneous. Further research for an association of clinical parameters and the patients' outcome is needed.

The study aims toward differences in the clinical and neurological outcome of surgical and non-surgical septic patients in comparison to non-septic patients on ICU. The aim of the study is to identify clinical and diagnostic outcome predictors in septic patients.

DETAILED DESCRIPTION:
All patients with severe sepsis and septic shock and fulfilling the inclusion criteria should be screened for the study on two surgical (septic surgical patients), one medical intensive care unit (septic non-surgical patients) and one neurological intensive care unit (non-septic patients) at the university hospital of Rostock, Germany.

The inclusion of patients will be started if written informed consent was obtained from all participants or their representatives (if direct consent could not be obtained).

The aim of the study is to determine differences in the neurological outcome of surgical and non-surgical septic patients (incidence, severity and length of critical-illness-polyneuropathy/-myopathy and septic encephalopathy). The main interest of the study is to find parameters associated with an improved neurological outcome in septic patients within an observation time of 100 days.

The main criterion is the incidence, severity and length of septic encephalopathy and critical-illness-polyneuropathy and -myopathy on days 7 and 28.

From all patients basic demographic data, illness severity scores (APACHE-II, SOFA) and delirium scores for the assessment of septic encephalopathy (CAM-ICU, ICDSC), laboratory, cerebrospinal fluid and microbiological results, electrophysiological (electroneurography(ENG)), electroencephalography (EEG), cranial MRI results, pre-morbidity data and clinical outcome for the study cohort will be recorded. At the days 1, 3, 7 and 28 the patients will be screened for clinical and laboratory/immunological data: hemodynamic, inflammation, coagulation, organ function, blood parameters including cytokines.

Neurological examination and EEG will be performed within 24 hours after the beginning of the study. Examination of liquor cerebrospinalis will be performed within 24-48 hours and cranial MRI between day 3 and 7 after the inclusion of the patient. ENG will be done earliest one week after the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling criteria for severe sepsis or septic shock

Exclusion Criteria:

* Diagnosis of cerebrovascular disease (pre-existing)
* Advanced dementia
* Diagnosis of pre-existing other neuromuscular disease
* High-dose glucocorticosteroid therapy (> 300 mg Hydrocortisone/die)
* Pre-existing renal replacement therapy
* Coagulation disorder with bleeding
* Frequent administration of neuromuscular blocking agents (> 3 times/week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with severe sepsis and septic shock and fulfilling the inclusion criteria should be screened for the study on two surgical (septic surgical patients), one medical intensive care unit (septic non-surgical patients) and one neurological intensive care unit (non-septic patients) at the university hospital of Rostock, Germany.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Septic Encephalopathy | day 7
  EEG, MRT, CSF (cerebrospinal fluid)
Critical-Illness-Polyneuropathy and -myopathy | day 7
  ENG
Septic Encephalopathy (28) | day 28
  Clinical observation.
Critical-Illness-Polyneuropathy and -myopathy (28) | day 28
  Clinical observation.

SECONDARY OUTCOMES:
- 28-day survival (observation time 100 days) | day 28
  Survival after 28 days.
- Time of respirator-therapy | 1 year
  In days cumulative.
- Dosage of vasopressors (cumulative) | observation time 100 days
  In days cumulative.
- 100 day survival | day 100
  Survival after 100 days.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, MD, Study Chair — University of Rostock
Locations (1):
- Intensive Care Units PIT 1+2, University hospital Rostock, Rostock, Germany

REFERENCES:
- [Derived] Ehler J, Barrett LK, Taylor V, Groves M, Scaravilli F, Wittstock M, Kolbaske S, Grossmann A, Henschel J, Gloger M, Sharshar T, Chretien F, Gray F, Noldge-Schomburg G, Singer M, Sauer M, Petzold A. Translational evidence for two distinct patterns of neuroaxonal injury in sepsis: a longitudinal, prospective translational study. Crit Care. 2017 Oct 23;21(1):262. doi: 10.1186/s13054-017-1850-7. PMID 29058589